CLINICAL TRIAL: NCT05770362
Title: Lifestyle Changes by the COVID-19 (Coronavirus Disease 2019) Pandemic in Children With Developmental Delays
Acronym: COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, MD, Professor, Taipei Medical University
Other Study IDs: MHW-111
Record Dates: First submitted 2023-03-10; First posted 2023-03-15 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Lifestyle-related Condition; COVID-19 Pandemic; Children With Developmental Delays
Keywords: COVID-19 pandemic; lifestyle; sleep; children with developmental delays
MeSH Terms: conditions — Mental Disorders; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: lifestyle questionnaire — The changes in lifestyle by lifestyle questionnaire during and after home isolation

SUMMARY:
To evaluate the lifestyle changes caused by the COVID-19 pandemic in children with developmental delays in Taiwan.

DETAILED DESCRIPTION:
Two hundred and sixty children with developmental delays in Shin Kong Wu Ho-Su Memorial Hospital will be included. The lifestyle questionnaire will evaluate the lifestyle changes of children with developmental delays during home isolation and release from home isolation during the COVID-19 pandemic in Taiwan. The parents of children with developmental delays will fill out the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* children diagnosed with developmental delays

Exclusion Criteria:

* children without developmental delays

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children diagnosed with developmental delays in Shin Kong Wu Ho-Su Memorial Hospital in Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2023-03-19 (Estimated); Primary Completion 2023-07-19 (Estimated); Study Completion 2023-07-19 (Estimated)

PRIMARY OUTCOMES:
sleeping quality change by lifestyle questionnaire | during and after home isolation through study completion, an average of 6 months
  Sleep quality changes during and after home isolation during the COVID-19 pandemic by lifestyle questionnaire. The minimum and maximum values range from 1 to 5; higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No